CLINICAL TRIAL: NCT00057408
Title: A Controlled Study of Olanzapine in Children With Autism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: FDA Office of Orphan Products Development (U.S. Federal Agency)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Richard P. Malone, MD, Drexel University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2190
Record Dates: First submitted 2003-04-01; First posted 2003-04-02 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2011-09

CONDITIONS: Autistic Disorder
Keywords: Autism; Pervasive Developmental Disorder; Treatment; Olanzapine; Antipsychotic
MeSH Terms: conditions — Autistic Disorder; Child Development Disorders, Pervasive | interventions — Olanzapine; Antipsychotic Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Treatment with olanzapine
  Interventions: Drug: olanzapine (Zyprexa)
- 2 (Placebo Comparator): Matching placebo treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: olanzapine (Zyprexa) — Olanzapine tablets given po at a dosage of 2.5 - 20 mg per day for up to 12 weeks.
  Other Names: Antipsychotic Drug
  Arms: 1
Drug: Placebo — Matching Placebo
  Other Names: Placebo controlled
  Arms: 2

SUMMARY:
This is a 12-week study which investigates the use of olanzapine to decrease disruptive behaviors sometimes associated with Autism in children, aged 3 to 12 years old. The first six weeks of the study are double-blind and placebo controlled, meaning that patients receive either placebo or olanzapine, and that neither the researchers nor the patients know whether or not they are receiving placebo or olanzapine. In the second six weeks all of the patients receive olanzapine. The purpose in using placebo is that it is otherwise impossible to know how effective the drug is or whether or not the drug causes side effects. Patients treated with placebo can have improvement and can have side effects. In the study patients receive a psychiatric evaluation, physical examination, laboratory tests, and study medication (olanzapine or placebo), free of charge.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, Aged between 3 and 12 years.
2. Autistic disorder - DSM-IV criteria.
3. A score of at least moderately impaired on the CGI-Severity item.
4. Clinical judgment that medication treatment for autism is indicated.

Exclusion Criteria:

1. Rett's disorder, childhood disintegrative disorder, Asperger's disorder, and PDD, NOS.
2. Psychotic disorder (DSM-IV) (including schizophreniform disorder and schizophrenia).
3. Major depressive disorder (DSM-IV).
4. Bipolar disorder (DSM-IV).
5. History of psychoactive drug in the previous 2 weeks prior to phase 1.
6. A history of treatment with olanzapine for a cumulative period of greater than 2 weeks prior to entering phase 1.
7. Systemic diseases such as cardiac, renal, thyroid diseases, uncontrolled seizure disorder (seizure disorder that is not controlled by anti-epileptic medication - a child who is seizure free for a period of 6 months on a stable dose of antiepileptic drug would be considered controlled), or diabetes mellitus.
8. Children with a known medical cause for autistic disorder.
9. Abnormal fasting blood glucose or history of diabetes.
10. Baseline body mass index (BMI) greater than the 90th percentile for age and gender (CDC growth charts, Kuczmarski et al, 2000) (because of risk of weight gain).
11. Baseline QTc >450 msec. Note: Historically, patients we evaluate do not have QTc values >450.
12. Dyskinesias at baseline (per the criteria of Schooler and Kane, 1982).

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Estimated)
Dates: Start 2003-05; Study Completion 2005-09

PRIMARY OUTCOMES:
Children's Psychiatric Rating Scale | Weekly

SECONDARY OUTCOMES:
Clinical Global Impressions | Weekly
Aberant Behavior Checklist | Weekly
Treatment Emergent Symptoms Scale | Weekly
Olanzapine Untoward Effects Checklist | Weekly
Abnormal Involuntary Movement Scale | Weekly
Neurological Rating Scale | Weekly

CONTACTS AND LOCATIONS:
Overall Officials: Richard P Malone, MD, Principal Investigator — Drexel University College of Medicine
Locations (1):
- Drexel University College of Medicine c/o Friends Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711